CLINICAL TRIAL: NCT01685177
Title: Prospective Randomized Trial Comparing Single-Anastomosis Duodeno-Ileal Bypass With Standard Roux-en-Y Duodenal Switch as a Second Step After a Sleeve Gastrectomy in the Super-Morbid Obese Patient
Brief Title: Single Anastomosis Duodeno-Ileal Bypass vs Standard Duodenal Switch as a Second Step After Sleeve Gastrectomy in the Super-Morbid Obese Patient
Acronym: SADI vs CD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Andres Sanchez-Pernaute, Chief, Esophago-Gastric and Morbid Obesity Surgery Unit, Hospital San Carlos, Madrid
Other Study IDs: SADI-CD
Record Dates: First submitted 2012-09-09; First posted 2012-09-14 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Morbid Obesity
Keywords: Morbid obesity; Sleeve gastrectomy; Duodenal Switch; SADI-S
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fat, liver tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SADI: Patients submitted to a second-step operation after a failed sleeve on which a single-anastomosis duodena-ileal bypass at 250 cm from the cecum is performed.

SUMMARY:
Single-Anastomosis Duodeno-Ileal bypass with a 250 cm common/alimentary loop is a modification of standard duodenal switch in which a Roux-en-Y duodeno-ileal anastomosis is performed at 250 cm from the cecum and a 60 cm to 100 cm common channel is build up. Hypothesis of the study is that Single-Anastomosis Duodeno-Ileal bypass behaves at least equally to standard duodenal switch as a second step after sleeve gastrectomy in the super-morbid patient. Secondary aims are to demonstrate that single-anastomosis duodeno-ileal bypass is simpler to perform, quicker and has less postoperative short, mid and long-term complications.

DETAILED DESCRIPTION:
Sleeve gastrectomy is a restrictive operation for morbid obesity which has a 60% success rate in solving both morbid obesity and related co-morbidities, mainly diabetes mellitus. When the sleeve is not enough for the patient, due to alimentary habits or to an excessive initial BMI before surgery (usually over 50 - 55), a second-step operation should be performed to increase effectiveness. Some patients are submitted to a second restrictive operation, i.e.: a re-sleeve, a gastric plication or sleeve banding. Other group are offered a gastric bypass. And, finally, a subset of patients, generally those with higher initial BMI, are offered a malabsorptive operation. While re-sleeve is adequate for many patients, gastric bypass is not offering a greater weight loss rate, and it is a complex operation requiring sectioning of the sleeve and two anastomoses. We support the performance of malabsorptive operations which warrant a better weight loss result for "resistant" patients needing a second-step. As Single-Anastomosis Duodeno-Ileal bypass with Sleeve gastrectomy (SADI-S) has behaved as a good primary operation for morbid obesity, we decided to test this one-loop reconstruction as a second step operation. Results will be compared to those obtained with a Roux-en-Y duodenal switch performed as a second step after a "failed" sleeve.

ELIGIBILITY:
Inclusion Criteria: Morbid obesity with initial BMI over 50 submitted to Sleeve Gastrectomy more than 18 months earlier. Excess weight loss with the sleeve under 50%.

-

Exclusion Criteria: Mental retard, alcoholism, age over 60, concomitant neoplastic disease.

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients attended in the Surgery Clinic with Morbid Obesity submitted to a sleeve gastrectomy and needing a second-step operation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-09

PRIMARY OUTCOMES:
Weight loss | 5 years from surgery
  Excess weight loss based on an ideal BMI = 25. EWL will be compared at 2 and 5 years from the second operation.

SECONDARY OUTCOMES:
Postoperative complications and nutritional complications | First 2 postoperative years
  Operative and postoperative complications (i.e.: leaks, bleeding, hernia...) will be recorded. Nutritional evolution (malnutrition) will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico San Carlos, Madrid, Madrid, Spain

REFERENCES:
- [Background] Sanchez-Pernaute A, Herrera MA, Perez-Aguirre ME, Talavera P, Cabrerizo L, Matia P, Diez-Valladares L, Barabash A, Martin-Antona E, Garcia-Botella A, Garcia-Almenta EM, Torres A. Single anastomosis duodeno-ileal bypass with sleeve gastrectomy (SADI-S). One to three-year follow-up. Obes Surg. 2010 Dec;20(12):1720-6. doi: 10.1007/s11695-010-0247-3. PMID 20798995
- [Background] Sanchez-Pernaute A, Rubio Herrera MA, Perez-Aguirre E, Garcia Perez JC, Cabrerizo L, Diez Valladares L, Fernandez C, Talavera P, Torres A. Proximal duodenal-ileal end-to-side bypass with sleeve gastrectomy: proposed technique. Obes Surg. 2007 Dec;17(12):1614-8. doi: 10.1007/s11695-007-9287-8. Epub 2007 Nov 27. PMID 18040751
- [Result] Sanchez-Pernaute A, Rubio MA, Perez Aguirre E, Barabash A, Cabrerizo L, Torres A. Single-anastomosis duodenoileal bypass with sleeve gastrectomy: metabolic improvement and weight loss in first 100 patients. Surg Obes Relat Dis. 2013 Sep-Oct;9(5):731-5. doi: 10.1016/j.soard.2012.07.018. Epub 2012 Aug 7. PMID 22963820